CLINICAL TRIAL: NCT02990572
Title: Research Contact Registry for Members of the Amish and Mennonite Communities
Brief Title: Amish/Mennonite Research Contact Registry
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Lina Ghaloul Gonzalez, Assistant Professor, Medical Genetics, University of Pittsburgh School of Medicine, University of Pittsburgh
Other Study IDs: STUDY20050302
Record Dates: First submitted 2016-11-30; First posted 2016-12-13 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: All
Keywords: Amish; Mennonite
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amish and Mennonite: * Agree to allow access to past, current, and future medical records
  * Provide a detailed family health history
  * Provide contact information that may be used for future approach regarding research studies

SUMMARY:
The purpose of this registry is to find members of the Plain Community who are interested in participating in future medical research studies. Having a registry makes it easier to contact and offer study participation to individuals who are appropriate for a new research study based on their own and their family medical history. Studies will focus on increasing knowledge about disorders affecting those who are Amish and Mennonite.

DETAILED DESCRIPTION:
The Amish and Mennonite communities of western Pennsylvania are unique because they are isolated both geographically and socially. These groups originally migrated as a small group from Europe. Since this first settlement there have been additional migration events within North America that have resulted in many distinct communities. These events lead to genetic founder effects, genetic bottleneck effects and virtually zero genetic inflow. The result has been an increased burden of genetic disease on these vulnerable communities. Specific founder genes explain the prevalence of different genetic conditions within each community and family group. This means that families and communities will have a clustering of certain genetic conditions, while the prevalence among the Plain people as a whole remains low. Understanding the specific needs of each family and community group is important in order to deliver comprehensive and specialized care. This requires research studies and needs assessments within these communities. Currently this need is being addressed in eastern Pennsylvania by the Clinic for Special Children in Strasburg. This organization has conducted research to improve access and quality of care for these Plain Communities. There is an apparent need for a similar understanding and relationship with the Plain Communities of western Pennsylvania.

Currently, a barrier exists for identifying and ascertaining appropriate individuals within the Plain Community for new research studies. This is largely due to their social and geographical isolation related to religious and cultural practices. Improving research and understanding within Plain Communities has the potential to improve early diagnosis, interventions, and clinical outcomes. Creating an ongoing registry will moderate these barriers and provide a platform for contacting willing members of the Plain Community for participation in future research projects that may positively impact their medical care, as well as the general care in their communities.

This is not a study but a registry. Potential participants will be educated about the intent of the registry, and written informed consent will be obtained to allow for collection and storage of information in the registry for an indefinite period of time. At the time of consent, potential participants will be informed about what it means to be a part of the registry and the potential for contact and recruitment to future research studies.

One-on-one interviews with a clinician, or with primary and co-investigators, will be conducted. This interview may take place in a clinic setting or the participants home or regional environment. The primary goal of the interview will be to collect a detailed family and medical history of each participant. This will be used to build a detailed pedigree of members of this community. Medical information obtained through released medical records will be included in the registry. Basic demographic and contact information will also be included in the registry.

Subjects information will be stored in the host PhenoTips database and data will be regularly undated and reviewed. Participants may be contacted for future research studies.

ELIGIBILITY:
Inclusion Criteria:

* Amish and Mennonite men and women age 18 or older
* Amish and Mennonite children with the permission of a parent

Exclusion Criteria:

* Amish and Mennonite men and woman age 18 or older who do not speak English
* Those who are not Amish or Mennonite

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Amish and Mennonite
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-10; Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Accumulation and clinical definition of a patient population who are willing to participate in future research studies for which they are eligible. | This registry is intended to be an ongoing resource for recruitment into future research studies and will be maintained up to 14 years.
  This research registry is intended to allow for identification of patients from the Plain Communities who are willing to participate in medical research. Eligibility for each future study will likely cary and patients will be selected and contacted with their permission, by dint of having consented to this registry, about the option of participating in a new research study.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Ghaloul Gonzalez, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No